CLINICAL TRIAL: NCT05577325
Title: The Effect Of Planned Educatıon Based On The Health Improvement Model On Lıfe Style Behavıors And Weıght Management In Obese Secondary School Students
Brief Title: The Effect Of Planned Educatıon Based On The Health Improvement Model
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Ayse Yilmaz (Other)
Responsible Party: Sponsor-Investigator, Ayse Yilmaz, lecturer/PhD student, Cumhuriyet University
Organization: Cumhuriyet University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ayse Yilmaz
Record Dates: First submitted 2022-04-25; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: OBESITY
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLANNED EDUCATION BASED ON THE HEALTH IMPROVEMENT MODEL (Experimental): Educational content based on the health promotion model, including nutrition and physical activity, will be created by the researcher by scanning the literature and considering the needs of the students. For the nutrition and physical activity plans included in the training, a diet specialist and a sports specialist will be consulted on the subject. The created training content and the booklet will be submitted to the opinion of at least three experts who are suitable for the subject area. Educational content deemed appropriate will be shared with students for 1 lesson per week for 10 weeks.
  Interventions: Behavioral: control group will be followed without health education
- follow without interference (Experimental): follow up without any education
  Interventions: Behavioral: control group will be followed without health education

INTERVENTIONS:
Behavioral: control group will be followed without health education — After the whole universe is evaluated in terms of percentile value, students with a percentile value of ≥95 will be filled with a pre-application form in terms of inclusion criteria in the research. Randomization will be made by drawing lots from the closed envelope in a way that will be homogeneously distributed between the classes and genders of the students who accept to participate in the research. Pre-tests will be given to those who accept to participate in the research. In the first week of the training, pedometers will be distributed and their use will be explained. This group is follow up without planned education. At the end of the sixth month of the study, the post-test data collection forms, excluding the personal information form, will be applied to the intervention group and anthropometric measurements will be made again.
  Other Names: Follow up without planned education

SUMMARY:
The aim of this study is to determine the effect of planned education based on the health promotion model on lifestyle behaviors and weight management in obese secondary school students.

DETAILED DESCRIPTION:
Obesity is a chronic disease that is explained by the increase in body fat mass compared to lean body mass, as a result of the fact that the energy taken into the body is more than the energy spent. Obesity, which is accepted as a complex and multifactorial disease that negatively affects health, is the second most important cause of preventable deaths after smoking. Obesity, cardiovascular diseases, especially type 2 diabetes and prediabetes, hypertension (HT), hyperlipidemia (HL), cerebrovascular disease, various cancers, obstructive sleep-apnea syndrome, non-alcoholic fatty liver disease, gastroesophageal reflux, biliary tract disease, It increases health expenditures by causing many health problems such as polycystic ovary syndrome, infertility, osteoarthrosis and depression.

Obesity is defined by the World Health Organization (2020) as "abnormal or excessive fat accumulation in the body to the extent that it impairs health". WHO (2020) reported that as of 2019, 38 million children under the age of 5 were overweight or obese in the world, and according to 2016 data, more than 340 million children and adolescents between the ages of 5-19 were overweight or obese. According to the results of Turkey Childhood Obesity Survey-2016, COSI-TUR (Childhood Obesity Surveillance Initiative), the rate of overweight in children aged 6-9 years was 14.6% and obesity rate was 9.9%. WHO (2016) reported that childhood obesity is one of the most serious public health problems of the 21st century, affecting many low- and middle-income countries, especially in urban environments, and that the problem is global.

With education becoming compulsory, schools are important places where children spend most of their lives independent of their families. In order for children to fully benefit from education, they must first be healthy. The age range of 6-12, also called school age, is stated as the period in which children's biopsychosocial development and growth is rapid, and they are most suitable for acquiring knowledge and gaining habits by gaining lifelong behaviors.

Although healthy, adequate and balanced nutrition is very important especially for children, as in all ages, it is known that nutritional problems are very common in this period. School-age children are among the groups most affected by inadequate and unbalanced nutrition. Another important problem accompanying the risk of unhealthy nutrition is the sedentary lifestyle. Technological factors (TV, internet), mostly driving to and from school, long working hours for exams, and unnecessary skipping of physical education classes lead children to a sedentary life. Children's adopting a more active lifestyle, increasing their physical activity levels and supporting them in this regard will make significant contributions to the social, mental and physical development of children.

The fact that childhood obesity is a global problem that seriously threatens public health brings forward initiatives to protect, which is the basis of the fight against obesity. Health professionals should ensure that children develop positive health behaviors and maintain these behaviors in adulthood by intervening on changeable factors such as lifestyle, nutritional behaviors and physical activity to prevent obesity. In order for the interventions to be successful, it is very important for health professionals to carry out their work in cooperation with parents, family and school.

Lifestyle changes and medical treatment are used in the treatment of obesity. In cases where lifestyle changes are unsuccessful, it is recommended to switch to medical treatment. On the other hand, it is stated that non-drug methods are very successful in improving mental health, quality of life and health, and are cost-effective in terms of not carrying risks and being inexpensive.

With the development of the nursing profession, the increase in its authority and responsibilities is closely related to the increase in its independent roles. One of the basic roles of the nurse is to provide education in a planned manner to protect and improve the health of the individual, family and society, to heal in case of illness and to gain the right health behaviors. Nursing knowledge is formed by nursing theories and conceptual models of nursing, and the new roles that have emerged in the nursing profession, nurses' other disciplines.

Unlike others, it requires the use of theories and models to improve care. Using nursing theoretical models in nursing practice provides a systematic approach to care and provides a scientific basis for practice-related concepts and principles. One of the most used models in the acquisition of health behaviors is the Health Promotion Model (SGM). SGM was developed by Pender between 1982-1984. The Health Promotion Model, which has features that will guide the practices related to health promotion, explains the factors that promote health and the factors that hinder it. In the model, factors that have direct and indirect effects on the health behavior of the individual are defined. According to Pender (1992), healthy lifestyle behaviors include spiritual development, health responsibility, exercise, nutrition, interpersonal relationships and stress management. The purpose of the model is to create a multivariate paradigm to explain and predict the components of lifestyle-related health promotion behaviors, to help nurses understand the determinants of healthy lifestyle behaviors, and to evaluate the individual's past life and other factors that may affect their perceptions of health behavior.

Eating healthy, maintaining a normal body weight, and coping with stress appropriately are stated as the key to achieving a healthy lifestyle for the individual. Obesity is closely related to the sub-dimensions of healthy lifestyle behaviors. Nutrition, physical activity and psychological factors are risk factors for obesity. Bad eating habits, sedentary life, increase in harmful habits cause the prevalence of obesity to increase day by day. Therefore, there is a strong relationship between the lifestyle habits of individuals and obesity. For this reason, it is recommended to monitor individuals with one or more risk factors for primary prevention, early detection of risks related to their lifestyle, and gaining healthy lifestyle behaviors to individuals. At this point, primary health care providers have important roles and responsibilities, and nurses are expected to support individuals in gaining healthy lifestyle behaviors.

The general goal in obesity management is to maintain or achieve normal BMI. The methods applied in the treatment of obesity can be grouped into five groups as Physical Activity, Behavioral Therapy, Nutritional Therapy, Medication, and Surgical Treatment. However, it is reported that it is inconvenient to apply drug therapy and surgical treatment in childhood, except in very compulsory situations. Studies on obesity indicate that nutritional therapy alone is not successful, that physical activity and nutrition therapy together provide more effective and long-term weight loss, and that lifestyle regulation and regular physical activity are essential to maintain weight loss. From this point of view, most of the programs to prevent obesity in children are about nutrition and physical activity. Changing individual behavior has been the main approach to prevent obesity. Schools are excellent learning environments for children. Most intervention studies on lifestyle and behavioral changes in children are school-based. School-based dietary and physical activity changes reduce the risk of obesity and chronic diseases and health expenditures . There are many examples of school-based nutrition and physical activity programs implemented in the world and in our country.

School health services carried out by the school health team are important in preventing obesity in children and protecting school children from obesity. Within the team that carries out school health services, the school health nurse has a key role in protecting and improving the health of students. Considering the role and responsibilities of the school nurse in eliminating the risk of obesity in school children; To prevent obesity, especially health education, to take health-promoting approaches, to determine risk groups by early diagnosis of overweight or obese children, to prevent the development of obesity in overweight children, to prevent the progression of obesity and the development of obesity-related complications in children who are determined to be obese. find it is clear that it is necessary. When nurses apply the necessary protection measures when they encounter children and families, the obesity rate and all risks that may develop due to obesity will be reduced. The purpose of this research; The aim of this study is to determine the effect of planned education based on the health promotion model on lifestyle behaviors and weight management in obese secondary school students.

ELIGIBILITY:
Inclusion Criteria:

* Being a middle school 6th and 7th grade student,
* Being ≥95 percentile according to percentile curves,
* Not having a chronic disease (metabolic syndrome, eating disorder, etc.) associated with obesity,
* Not using drugs continuously
* Not having a physical disability to be able to do physical activity,
* Not having a mental disability.

Exclusion Criteria:

* Although they have accepted to participate in the research those who want to quit the study voluntarily during the research process,
* Do not participate in the trainings and counseling programs given within the specified time period,
* And are diagnosed with any health problem,

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 112 (Estimated)
Dates: Start 2022-01-13 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
nutritional self-efficacy | 12 weeks
  increase in nutritional self-efficacy scores
physical activity | 12 weeks
  increased physical activity scores
lifestyle behavior | 24 weeks
  increase in lifestyle behavior scores
percentile-BMI values | 18 weeks
  normal percentile-BMI values

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Yilmaz, Principal Investigator — Cumhuriyet University; Semra Zorlu, Principal Investigator — Cumhuriyet University
Locations (2):
- Turkey (Türkiye) (2):
  - Mevlana Vali Zubeyir Kemelek Secondary School, Sivas
  - Selcuk Secondary School, Sivas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alıcı, M., Pınar, R. (2008). Obez hastalara verilen eğitimin etkinliğinin değerlendirilmesi. Hemşirelikte Araştırma Geliştirme Dergisi, 2: 32-47.
- [Background] Appleton J, Fowler C, Brown N. Parents' views on childhood obesity: qualitative analysis of discussion board postings. Contemp Nurse. 2017 Aug;53(4):410-420. doi: 10.1080/10376178.2017.1358650. Epub 2017 Aug 1. PMID 28728473
- [Background] Bahar, Z. (2010). Okul Sağlığı Hemşireliği. Dokuz Eylül Üniversitesi Hemşirelik Yüksekokulu Elektronik Dergisi, 3 (4):195-200.
- [Background] Bahar. Z., Açıl. D. (2014) Sağlığı Geliştirme Modeli: Kavramsal Yapı. Dokuz Eylül Üniversitesi Hemşirelik Yüksekokulu Elektronik Dergisi 7 (1).ss: 59-67
- [Background] Bayazıt Hayta, A., Şanlıer, N.(2007). İlköğretim 6. 7. 8. Sınıf Öğrencilerinin Beslenme Davranışları Ve Sosyal Onaylanma İsteği. Milli Eğitim Dergisi, 174.
- [Background] Berberoğlu M. (2008). Adölesanlarda obezite. İ. Ü. Cerrahpaşa Tıp Fakültesi Sürekli Tıp Eğitimi Etkinlikleri Adolesan Sağlığı II Sempozyum Dizisi, 63: 79- 80.
- [Background] Bilici, S., Köksal, E.(2013). Okul Öncesi ve Okul Çağı Çocuklara Yönelik Beslenme Önerileri ve Menü Programları. Şanlıer, N.(Ed). Sağlık Bakanlığı Yayınları, Ankara.
- [Background] COSI-TUR (2017). Türkiye Çocukluk Çağı (İlkokul 2. Sınıf Öğrencilerde) Şişmanlık Araştırması Cosı-Tur 2016. Sağlık Bakanlığı Yayın No:1080, Ankara.
- [Background] Iversen CS, Nigg C, Titchenal CA. The impact of an elementary after-school nutrition and physical activity program on children's fruit and vegetable intake, physical activity, and body mass index: Fun 5. Hawaii Med J. 2011 Jul;70(7 Suppl 1):37-41. PMID 21886292
- [Background] Ergül, Ş., Kalkım, A. (2011). Önemli Bir Kronik Hastalık: Çocukluk ve Ergenlik Döneminde Obezite. TAF Preventive Medicine Bulletin, 10(2): 223-230.
- [Background] Kriemler S, Zahner L, Schindler C, Meyer U, Hartmann T, Hebestreit H, Brunner-La Rocca HP, van Mechelen W, Puder JJ. Effect of school based physical activity programme (KISS) on fitness and adiposity in primary schoolchildren: cluster randomised controlled trial. BMJ. 2010 Feb 23;340:c785. doi: 10.1136/bmj.c785. PMID 20179126
- [Background] Meydanlıoğlu A. (2013) Hemşire Liderli Sağlik İçin Beslenme ve Fiziksel Aktivite Programi'nın Çocuklarin Beslenme ve Fiziksel Aktivite Düzeylerine Etkisi. Yayınlanmış Doktora Tezi, Marmara Ü. SBE, Halk Sağlığı Hemşireliği ABD.
- [Background] Neumark-Sztainer D, Story M, Hannan PJ, Rex J. New Moves: a school-based obesity prevention program for adolescent girls. Prev Med. 2003 Jul;37(1):41-51. doi: 10.1016/s0091-7435(03)00057-4. PMID 12799128
- [Background] Pender, N.J., Murdaugh, C.L. ve Parsons, M.A. (2002) Health Promotion in Nursing Practice, Fourth Edition, New Jersey, 13-209.
- [Background] Pyle, S., Sharkey, J., Yetter, G., Felıx,E., Furlong, Mj.(2006). Fıghtıng An Epıdemıc: The Role Of Schools In Reducıng Chıldhood Obesıty. Psychology in the Schools, 43(3): 361-376.
- [Background] Udemgba C, Sharma M. (2015). ChildhoodObesity: A QualitativeReview of School-BasedInterventions. Austin J Obes&MetabSynd. 1(1): 1004.
- [Background] Martinez Vizcaino V, Salcedo Aguilar F, Franquelo Gutierrez R, Solera Martinez M, Sanchez Lopez M, Serrano Martinez S, Lopez Garcia E, Rodriguez Artalejo F. Assessment of an after-school physical activity program to prevent obesity among 9- to 10-year-old children: a cluster randomized trial. Int J Obes (Lond). 2008 Jan;32(1):12-22. doi: 10.1038/sj.ijo.0803738. Epub 2007 Sep 25. PMID 17895883
- [Background] Yabancı N. (2011) Okul sağlığı ve beslenme programları. TAF Preventive Medicine Bulltein;10(3):361-368.
- See also: Related Info — http://www.who.int/news-room/fact-sheets/detail/obesity-and-overweight
- See also: Related Info — http://www.cdc.gov/nchs/data/databriefs/db288.pdf

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-01-13): https://cdn.clinicaltrials.gov/large-docs/25/NCT05577325/Prot_SAP_ICF_000.pdf